CLINICAL TRIAL: NCT05496400
Title: Effect of Anemia of Prematurity and Its Treatment on Hemodynamics of Preterm Infants
Brief Title: Anemia of Prematurity and Hemodynamics
Status: Completed | Type: Observational
Sponsor: Marwa Mohamed Farag (Other)
Responsible Party: Sponsor-Investigator, Marwa Mohamed Farag, Primary Investigator and Lecturer in Pediatrics, Faculty of Medicine, Alexandria University
Organization: Alexandria University (Other)
Other Study IDs: 0106769
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: (anemic group)
  Interventions: Radiation: Echocardiographic and Doppler studies
- Group II: (non-anemic group)
  Interventions: Radiation: Echocardiographic and Doppler studies

INTERVENTIONS:
Radiation: Echocardiographic and Doppler studies — Echographic and Doppler studies will be performed using machine: model GE Vivid iq premium,WUXI,China and we will measure:
  1. Cardiac output:
  2. Cerebral, intestinal and renal blood flow velocities:

SUMMARY:
The aim of this work to study the hemodynamic changes accompanying anemia of prematurity in neonates with gestational age ≤32 weeks and the effect of its treatment on hemodynamics.

DETAILED DESCRIPTION:
This prospective observational study aims to evaluate the hemodynamic changes provoked by anemia of prematurity and transfusion of packed red blood cells (RBCs). Nonanemic inpatient premature infants (Hematocrit>30%) will be compared with pretransfusional anemic inpatient premature infants. Anemic premature infants will be assessed before and 24 hours after the transfusion of pRBCs. Cerebral, intestinal and renal blood flow velocities, cardiac output parameters will be measured in premature neonates who will fulfill the eligibility criteria of the study.This study will be conducted at the neonatal intensive care units in Alexandria University Hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants ≤32 weeks gestational age, regardless their weight with postnatal age 3-6 weeks.

Exclusion Criteria:

-

Ages: 3 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients with any of the following will be excluded at the time of assessment:
  * Hemolytic disease of the newborn.
  * Shock.
  * Sepsis.
  * Ultrasonographic abnormalities of kidney, heart and cerebral structures.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
1. Cardiac output: | 3-6 weeks postnatal age
  Probe: GE 12S-RS probe with a frequency range of 5 - 11 MHz. Cardiac output as the product of stroke volume and heart rate: actual body weight in mL/kg/min; Stroke volume (the product of velocity time integral at the level of aortic valve pulsed wave (PW) and cross-sectional area of the left ventricular outflow tract at the level of aortic valve using 2D.(
2. Cerebral blood flow velocities | 3-6 weeks postnatal age
  in the anterior cerebral artery through the anterior fontanelle in the sagittal plane
3. Intestinal blood flow velocities | 3-6 weeks postnatal age
  in the celiac artery from a longitudinal abdominal section, determined close to the origin of the artery from the abdominal aorta.
4.Renal blood flow velocities | 3-6 weeks postnatal age
  Renal blood flow velocities in the right renal artery by placing the transducer below the right costal arch in the dorsolateral area of the flank in longitudinal axis.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Adel El Beheiry, PhD, Study Chair — Faculty of medicine, Alexandria University, Egypt; Amany Tolba Elsebaee, MBBCh, Principal Investigator — Faculty of medicine, Alexandria University, Egypt
Locations (1):
- Neonatal Intensive Care Unit (NICU) of Alexandria University Maternity Hospital., Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided